CLINICAL TRIAL: NCT03962296
Title: A Multicenter, Randomized, Double-blind Non-inferiority Trial to Evaluate the Efficacy and Safety of Entelon® as Compared to Doxium Tab. And Placebo for the Treatment of Nonproliferative Diabetic Retinopathy
Brief Title: A Multicenter, Randomized, Double-blind Non-inferiority Trial to Evaluate the Efficacy and Safety of Entelon®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanyang University (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Un shin, Investigator, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENTL_501
Record Dates: First submitted 2019-05-16; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic retinopathy, hard exudates
MeSH Terms: conditions — Diabetic Retinopathy | interventions — whole grape extract; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Entelon (Experimental): Three daily oral doses of 50mg tablets were administered to patients
  Interventions: Drug: Vitis vinifera extract
- Doxium (Active Comparator): Three daily oral doses of 250mg tablets were administered to patients
  Interventions: Drug: Calcium Dobesilate
- Placebo (Placebo Comparator): Three masking tablets were administered to patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitis vinifera extract — Three daily oral doses of 50mg tablets of Vitis vinifera extract(Entelon®, Hanlim Pharm, Seoul, South Korea) were administered to patients in this group
  Other Names: Experimental: Entelon
  Arms: Entelon
Drug: Calcium Dobesilate — Three daily oral doses of 50mg tablets of Calcium Dobesilate(Doxium®, Ilsung Pharm, Seoul, South Korea) were administered to patients in this group
  Other Names: Active comparator:Doxium
  Arms: Doxium
Drug: Placebo — Placebo tablets lacked Vitis vinifera extract or calcium dobesilate, but their appearance was identical to those of the study group tablets.
  Other Names: Placebo comparator:Placebo
  Arms: Placebo

SUMMARY:
This was a multicentre, randomised, double-blind controlled study that compared the efficacy and safety of V. vinifera extract, calcium dobesilate (CD), and placebo in subjects with DME. Patients made 6 clinic visits, namely the screening visit; baseline visit (T0); and follow-up visits at 3 (T3), 6 (T6), 9 (T9), and 12 (T12) months.

DETAILED DESCRIPTION:
Eligible patients were randomised to one of the three study groups in a 1:2:2 ratio (placebo:GSPE:CD group). The randomization schedule was generated and prepared using cubeIWRS® solution (CRScube Inc., Seoul, South Korea, HQ). Randomization was performed using a complete randomization algorithm according to the order of the baseline visit. Subjects took three tablets of a masked study medication three times daily for 12 months; the first dose was taken in the morning of the baseline visit (T0) after baseline assessments were performed, and the last dose was taken in the evening before the month 12 visit (T12). Three daily oral doses of 50mg tablets of GSPE (Entelon®, Hanlim Pharm, Seoul, South Korea) were administered to patients in the GSPE group. Placebo tablets lacked GSPE, but their appearance was identical to that of the study group tablets. Commercially available 250mg CD tablets (Doxium®, Ilsung Pharm, Seoul, South Korea) were used in this study. The identity of the masked study medications was concealed by storing the medications in individually sealed envelopes at the study sites.

ELIGIBILITY:
Inclusion Criteria:

* Singing a written informed consent prior to selection
* type 2 DM aged between 40 and 80 years
* Diabetes is well controlled with drugs for at least 3 months(HbA1c ≤9%)
* Best-corrected visual acuity over 0.5(20/40) by using ETDRS cisual acuity test
* Diabetic macular edema with hard exudates CSMT ≤300µm

Exclusion Criteria:

* Lase therapy or intravitreal injection(anti-VEGF, steroid) intraocular surgery within 6 months of enrollment
* Concomitant macular disease (such as retinal vascular occlusion, choroidal neovascularization, epiretinal membrane, etc)
* Poor image of optical coherence tomography(signal strength under 50% of narmal value)
* Concomitant therapy(Kallidinogenase, Vaccinium myrtillus extract, sulodexide)
* Non-controlled hypertension(systolic pressure >140mmHg or diastolic pressure <90mmHg)
* Severe renal insufficiency(creatinine >2.2mg/dL, or undergoing dialysis)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2015-01-26 (Actual); Study Completion 2015-01-26 (Actual)

PRIMARY OUTCOMES:
The change(Improvement)in the hard exduates | T0(baseline), T12(12months)
  The improvement of HE was defined as a decrease in the HE severity by at least two categories of severity at T12 compared with the baseline visit.

SECONDARY OUTCOMES:
The change of Best-corrected visual acuity(BCVA) | T0(baseline), T3(3months), T6(6months), T9(9months), T12(12months)
  Using the Early Treatment Diabetic Retinopathy Study(ETDRS) protocol
The change of central subfield mean thickness(CSMT) | T0(baseline), T3(3months), T6(6months), T9(9months), T12(12months)
  Using 6-radial scan protocol or cube scan protocol according to local guidelines of each center;the ETDRS style map
The change of total macular volum(TMV) | T0(baseline), T3(3months), T6(6months), T9(9months), T12(12months)
  Using 6-radial scan protocol or cube scan protocol according to local guidelines of each center;the ETDRS style map

CONTACTS AND LOCATIONS:
Overall Officials: Ha kyoung Kim, PhD, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spadea L, Balestrazzi E. Treatment of vascular retinopathies with Pycnogenol. Phytother Res. 2001 May;15(3):219-23. doi: 10.1002/ptr.853. PMID 11351356